CLINICAL TRIAL: NCT06849635
Title: Cera™ ASD Occluder Post-Market Clinical Follow-Up Study：A Multi-Center, Single-arm, Ambispective Post-Market Follow-Up Study
Brief Title: Cera™ ASD Occluder Post-Market Clinical Follow-Up Study
Status: Recruiting | Type: Observational
Sponsor: Lifetech Scientific (Shenzhen) Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: LT-TS-27-2025-01
Record Dates: First submitted 2025-02-08; First posted 2025-02-27 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Atrial Septal Defect
Keywords: Atrial Septal Defect
MeSH Terms: conditions — Heart Septal Defects, Atrial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this post-market study is to:

* collect real-word clinical data and confirm the long-time safety and performance of the Lifetech Cera™ ASD Occluder
* identify previously unknown side-effects

DETAILED DESCRIPTION:
Atrial Septal Defect (ASD) is a type of Congenital Heart Defects (CHD) that have the potential to be closed without open-heart surgery. The treatment of choice for ASD closure has long been surgical closure. An alternative is the use of percutaneous access and transcatheter occluder devices as a treatment option for ASD. With percutaneous closure a thoracotomy is no longer needed and this is associated with a decreased procedural time and shorter hospital stay. The Lifetech Cera™ ASD occluder is a percutaneous, transcatheter closure device for the non-surgical closure of ASD. In order to collect real-word clinical data and confirm the long-time safety and performance of the Lifetech Cera™ ASD Occluder, this post-market clinical follow-up study is planned under the Regulation (EU) 2017/745. The study intends to enroll 139 subjects. The anticipated enrollment period is approximately 1 years and subjects will be followed for 2 years (24 months) post-implantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of secundum Atrial Septal Defect (ASD).
* Patients was implanted with the study device from 01 Jan 2020 to 31 Dec 2023 as per IFU instructions.
* Patients or legally authorized representative are willing to the collection and processing of his/her data or sign the Informed Consent.

Exclusion Criteria:

* Patients who have extensive congenital cardiac anomaly which can only be adequately repaired by cardiac surgery.
* Patients who have sepsis within one month prior to implantation, or any systemic infection that can't be successfully treated prior to device placement.
* Patients known to have a bleeding disorder, untreated ulcer or any other contraindications to aspirin therapy, unless another anti-platelet agent can be administered for 6 months.
* Patients who have demonstrated intra-cardiac thrombi on echocardiography (especially left atrial or left atrial appendage thrombi).
* Patients whose size (i.e., too small to tolerate TEE probe, catheter size, etc.) or condition (active infection, etc.) would cause the patient to be a poor candidate for cardiac catheterization.
* Patients where the margins of the defect are less than 5mm from the coronary sinus, AV valves or right upper lobe pulmonary vein.
* Patients did not conduct any follow up visit after hospital discharge.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a confirmed diagnosis of secundum Atrial Septal Defect (ASD), who needs endovascular aortic repair.
Sampling Method: Probability Sample
Enrollment: 139 (Estimated)
Dates: Start 2025-01-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Procedural success | 6 months post-implantation
  1. Absence of stroke/TIA, device embolization, cardiac or vascular perforation or device/procedure related death, assessed at 6 months post-implantation.
  2. Successful closure of the defects, with no, trivial or small residual shunt confirmed by Doppler echocardiography at 6 months post-implantation.

SECONDARY OUTCOMES:
Successful closure of the defects | at procedure, discharge（up to 2 days）and 12 months post-implantation
  With no, trivial or small residual shunt confirmed by Doppler echocardiography
Incidence of new onset arrhythmia requiring medical treatment | From attempted procedure to 2 years post-implantation
  Include medication, intervention or surgical treatment
Incidence of device or procedure related Adverse Events (AEs) | From attempted procedure to 2 years post-implantation
  Untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the study medical device and whether anticipated or unanticipated.
Incidence of device or procedure related Serious Adverse Events (SAEs) | From attempted procedure to 2 years post-implantation
  Adverse event that led to any of the following:
  1. death,
  2. serious deterioration in the health of the subject, users, or other persons as defined by one or more of the following:
     1. a life-threatening illness or injury, or
     2. a permanent impairment of a body structure or a body function including chronic diseases, or
     3. in-patient or prolonged hospitalization, or
     4. medical or surgical intervention to prevent life-threatening illness or injury, or permanent impairment to a body structure or a body function,
  3. foetal distress, foetal death, a congenital abnormality, or birth defect including physical or mental impairment
Incidence of death | From attempted procedure to 2 years post-implantation
  Death

CONTACTS AND LOCATIONS:
Locations (6):
- Poland (6):
  - G.V.M.Carint Hospital, Myszków
  - Centre for Invasive Cardiology, Electrotherapy and Angiology G.V.M.Carint-Oswiecim, Oświęcim
  - Subcarpathian Centre for Cardiovascular Intervention G.V.M.Carint -Sanok, Sanok
  - Polish-American Heart Clinics, Heart and Vascular Center in Tychy, American Heart of Poland Group, Tychy
  - Polish-American Heart Clinics 1st Department of Invasive Cardiology and Heart Failure in Ustroń, AHoP Group, Ustroń
  - Dr. Tytus Chałubiński County Hospital, Zakopane